CLINICAL TRIAL: NCT05207631
Title: Misused Inhaler and Insufficient Peak Inspiratory Flow in Hospitalized COPD Patients Before and After Implementation of a Systematic Assessment and a Prescription Guide - a Quasi Experimental Study - MIPIF
Brief Title: Intervention to Reduce Misused Inhaler and Insufficient Peak Inspiratory Flow in Hospitalized COPD Patients
Acronym: MIPIF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital Fribourgeois (Other)
Responsible Party: Principal Investigator, Gaël Grandmaison, Doctor, Hôpital Fribourgeois
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 010322
Record Dates: First submitted 2021-12-29; First posted 2022-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: COPD
Keywords: Inhaler; Critical error; Inspiratory peak flow; Hospital
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Quasi-experimental study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control cohort (No Intervention): Participants in the control cohort received standard care.
- Cohort with intervention (Active Comparator): Participants included in the intervention cohort receive a systematic and standardised assessment of their inhaler on admission to our department. Their inhalers are adapted in accordance with a prescribing guide.
  Interventions: Other: Systematic and standardised assessment of inhalers and implementation of a prescribing guide

INTERVENTIONS:
Other: Systematic and standardised assessment of inhalers and implementation of a prescribing guide — Participants included in the intervention cohort receive a systematic and standardised assessment of their inhalers on admission to our department. The assessment is carried out by a physiotherapist and aims to assess inhalation technique, peak inspiratory flow and ability to use the inhaler after targeted teaching. Based on this information and a prescription guide provided, the patient's doctor can select the most appropriate inhaler.
  Arms: Cohort with intervention

SUMMARY:
The drug treatment of chronic obstructive pulmonary disease (COPD) is mainly based on inhaled therapy. This route of administration is limited by inhaler handling errors, insufficient inspiratory flow or inappropriate inhalers. According to the scientific literature, these limitations are extremely common in both outpatients and inpatients.

Our hypothesis is that the implementation of a standardised and systematic assessment of inhalers combined with a prescribing guide to help select a suitable inhaler will decrease the proportion of suboptimally used inhalers at discharge in patients hospitalised with a diagnosis of COPD.

To assess the effectiveness of our intervention, the investigators will compare the proportion of inhalers used suboptimally at hospital discharge between a control cohort before the implementation of our intervention and a cohort after the implementation of our intervention. Secondary outcomes include reasons for sub-optimal use of inhalers, i.e. inhaler handling errors, insufficient peak inspiratory flow or inappropriate inhaler. Secondary outcomes will also include length of hospital stay and 30-day readmission rate.

ELIGIBILITY:
Inclusion Criteria:

1. Admission to the HFR Fribourg internal medicine department
2. Age greater than or equal to 18 years
3. Diagnosis of COPD
4. Use of an inhaler device for the treatment of COPD before admission

Exclusion Criteria:

1. Inability to complete initial assessment due to language problems
2. Inability to complete initial assessment due to physical or mental conditions
3. Patient who has already received the intervention during a previous hospitalization.
4. Length of hospitalization of less than 72 hours
5. Patient already included in the control period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-12-25 (Actual); Study Completion 2023-01-24 (Actual)

PRIMARY OUTCOMES:
Proportion of inhalers used sub-optimally at hospital discharge | This outcome is assessed within 48 hours prior to hospital discharge
  An inhaler used sub-optimally is defined as an inhaler used with at least one critical error and/or with insufficient inspiratory flow.

SECONDARY OUTCOMES:
Proportion of inhaler used with a critical error at hospital discharge | This outcome is assessed within 48 hours prior to hospital discharge
  In accordance with the literature, the investigators define critical error as an action or an inaction that in itself would have a detrimental impact of the delivery of the drug to the distal airways.
Proportion of inhaler used with suboptimal peak inspiratory flow at hospital discharge. | This outcome is assessed within 48 hours prior to hospital discharge
  The peak inspiratory flow values considered sub-optimal for inhaler use are defined in the literature and are specific to each inhaler type.
Proportion of inhalers that cannot be handled properly despite appropriate teaching at hospital discharge. | This outcome is assessed within 48 hours prior to hospital discharge
  If critical errors are identified in the handling of the inhaler, the physiotherapist provides targeted instruction to correct these errors. After each instruction, a new assessment of the inhaler technique is performed and the instruction is repeated if a critical error persists. If handling critical errors persist despite appropriate instruction, it's considered that the inhaler cannot be handled by the patient.
Proportion of inappropriate inhaler at hospital discharge. | This outcome is assessed within 48 hours prior to hospital discharge
  An inhaler is considered unsuitable if the patient is unable to handle it properly after appropriate instruction and/or if the patient does not have sufficient inspiratory flow for optimal use of the inhaler.
Proportion of inhalers used sub-optimally at hospital discharge by type of inhaler. | This outcome is assessed within 48 hours prior to hospital discharge
  The proportion of inhalers used sub-optimally at hospital discharge is described by type of inhaler.
Proportion of patients using at least one inhaler sub-optimally | This outcome is assessed within 48 hours prior to hospital discharge
  A participant is considered to have suboptimal device use if making a critical error when using an inhaler or if their peak inspiratory flow rate is insufficient for optimal device use.
Length of hospital stay | This outcome is assessed up to three months
  The length of stay in acute care on the internal medicine department will be documented.

CONTACTS AND LOCATIONS:
Overall Officials: Gaël Grandmaison, Dr, Principal Investigator — Hôpital Fribourgeois
Locations (1):
- HFR Fribourg, Fribourg, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grandmaison G, Grobety T, Dumont P, Vaucher J, Hayoz D, Suter P. An in-hospital intervention to reduce the proportion of misused inhalers at hospital discharge among patients with COPD: a non-randomised intervention study. Swiss Med Wkly. 2024 Apr 4;154:3394. doi: 10.57187/s.3394. PMID 38579300